CLINICAL TRIAL: NCT03197948
Title: A Pilot Feasibility Trial Examining the Use of Electronic Patient-Reported Outcomes in Prostate Cancer Patients With Apple ResearchKit Smartphone Application
Brief Title: Electronic Patient Reported Outcomes in Measuring Health-Related Quality of Life in Patients With Stage I-IV Prostate Cancer Undergoing Treatment
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 16G.052; JT 8603 (Other: JeffTrial Number)
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Services Research (electronic patient reported outcome): Patients complete questionnaires over 15 minutes once a week over 3 months via a smartphone application. Patients rate urinary function, bowel habits, sexual function, hormonal function, and overall satisfaction. Patients with advanced disease also answer questions related to pain, fatigue/lack of energy, weight loss, and worry domains.
  Interventions: Other: Internet-Based Intervention

INTERVENTIONS:
Other: Internet-Based Intervention — Complete questionnaire via a smartphone application

SUMMARY:
This pilot clinical trial studies how well electronic patient reported outcomes work in measuring health-related quality of life in patients with stage I-IV prostate cancer undergoing treatment. Using a smartphone application to measure and monitor symptoms before, during, and after treatment may help patients better detect, understand, and manage their health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the feasibility of collecting electronic patient-reported outcome data using validated health-related quality of life (HRQOL) assessment tools at baseline, during, and after treatment through a smartphone application in adult men throughout their course of treatment for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported ability to speak and read English
* Be able to communicate on a touch screen iPhone
* Willing to provide signed informed consent
* Willing and able to comply with all study activities
* Access to WiFi connection or cellular data
* An established clinical history of prostate cancer in a spectrum of severity (all stages)

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if in the investigator's opinion the patient has any concurrent medical or psychiatric condition that may preclude participation in this study or completion of self-administered questionnaires (e.g., moderate to severe dementia and/or severe, uncontrolled schizophrenia, or other condition that would render them unable to complete a questionnaire)
* Cognitive or other impairment (e.g., visual) that would interfere with completing a self- administered questionnaire and with participating in a group discussion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will consist of adult male volunteers, all of whom will be participating in a prostate cancer treatment clinical trial at Thomas Jefferson University Sidney Kimmel Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Feasibility defined as satisfactory completion (60%) of weekly questionnaires | Up to 3 months
  The rate of satisfactory completion will be estimated along with a one-sided exact 95% confidence interval. The method will be considered feasible if the lower bound of the confidence interval is above 0.7 or, equivalently, if at least 49/60 (82%) of participants have satisfactory completion. Rates of completion may be estimated by levels of baseline demographic or clinical characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dicker, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/